CLINICAL TRIAL: NCT02859792
Title: Riluzole in the Treatment of Spasticity in the Traumatic Chronic Spinal Cord Injury Condition: Adaptive, Multicenter, Placebo-controlled, Randomised, Double Blind Trial in a Rare Disorder
Brief Title: Riluzole in the Treatment of Spasticity in the Traumatic Chronic Spinal Cord Injury Condition
Acronym: RILUSCI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-000901-35; 2016-02 (Other: ap hm)
Record Dates: First submitted 2016-08-02; First posted 2016-08-09 (Estimated); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Riluzole; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Biological: Blood Samples
- Experimental (Experimental)
  Interventions: Drug: Riluzole; Biological: Blood Samples

INTERVENTIONS:
Drug: Riluzole — Riluzole capsules (25 or 50 mg) will be administered in the four dose level groups (i.e. 25 mg bid; 50 mg bid; 75 mg bid; 100 mg bid).
  Arms: Experimental
Drug: Placebo — placebo capsules 25 or 50 mg
  Arms: Placebo
Biological: Blood Samples — v1;v2;v3;v4

SUMMARY:
The study will be conducted in two steps:

1. Determination of the Minimal Effective Dose (MED) among the four doses of the panel
2. Estimation of the probability of response associated to the MED.

Each step has a main objective:

Step 1 Objective: To determine a daily dose of Riluzole that improves spasticity in patients with chronic SCI

Step 2 Objective: To demonstrate, in a phase 2b trial, the efficacy of Riluzole to improve spasticity vs placebo, in patients with chronic SCI.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic traumatic SCI defined as:

   a. At least a 12-month history of:

   i. C4-T12 traumatic SCI

   ii. Complete and incomplete ( AIS A,B,C,D)

   iii. With Spasticity (5>MAS>1 on at least adductor muscles and/or triceps surae muscles and NRS ≥ 4)
2. Male or Female
3. Aged 18 to 65 years at the time of screening
4. Judged by site investigator to be able to comply with evaluations at baseline and throughout the study
5. Last injection of BTX-A in striated muscle more than 3 months ago and patients must have returned to their level of spasticity before BTX-A injection
6. Last intrathecal (IT) injection of baclofen or per os administration of any myorelaxant should be more than 14 days ago (Step 1)
7. The dose of myorelaxant or Baclofen should be stable for ≥ 30 days prior to screening and kept at stable daily dose until the end of the protocol (Step 2).
8. Stable on all other chronic medications for ≥ 30 days prior to screening, including analgesics
9. Stable on rehabilitation (methods and frequency) for ≥ 15 days prior to screening
10. Written informed consent provided by subject

Exclusion Criteria:

1. Spinal cord injury of less than 12 months,
2. Associated Brain lesion that might be the cause of spasticity,
3. MAS≤1 or =5 on at least adductor muscles and/or triceps surae muscles or NRS < 4
4. Presence of urinary infection, fever, pressure ulcer or other spasticity-aggravating factors.
5. Presence of other significant neurological or mental disorder or other illness, which would preclude accurate evaluation,
6. Recent history (less than 1 year) of chemical substance dependency or significant psychosocial disturbance,
7. Insufficient fluency in local language to complete neuropsychological, global and spasticity assessments
8. Active liver disease or clinical jaundice
9. Active malignancy or history of invasive malignancy within the last five years
10. Neutropenia, liver enzymes (ALT/SGPT or AST/SGOT) 2 times the upper limit of normal (ULN) at screening visit, baseline elevations of several liver function tests (especially elevated bilirubin).
11. AIDS or AIDS-related complex,
12. The systolic blood pressure measurement is > 190 or < 85 mm Hg and/or the diastolic blood pressure measurement is > 105 or < 50 mm Hg at screening.
13. The ECG is abnormal at screening and judged to be clinically significant by the site investigator. Particular attention will be given to any sign suggesting conduction disorders.
14. Treatment with any investigational drugs or device within 60 days of screening
15. Any myorelaxant medication including IT baclofen, taken by the subject in the last 14 days prior to screening (step 1)
16. Not stable under IT baclofen or per os myorelaxant medication for at least 30 days prior screening (step 2)
17. Not stable on all other chronic medications for ≥ 30 days prior to screening, including analgesics
18. Injection of BTX-A in striated muscle less than 3 months ago
19. Subject is currently using, and will continue to use for the next 14 days any of the following medications which are classified as Inhibitors of CYP 1A2 (e.g. diclofenac, diazepam, nicergoline, clomipramine, imipramine, fluvoxamine, phenacetin, theophylline, amitriptyline and quinolones) or Inducers of CYP 1A2 (e.g. rifampicin and omeprazole)
20. Ongoing pregnancy or lactation. Women with childbearing potential not using any form of efficacious contraception.
21. Known hypersensitivity to Riluzole

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-05-27 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
the Minimum Effective Dose (MED) of Riluzole | 2 Months
  Blood Sample

CONTACTS AND LOCATIONS:
Overall Officials: Catherine GEINDRE, Study Director — Assistance Publique Hopitaux De Marseille; OLIVIER BLIN, Principal Investigator — Assistance Publique Hopitaux De Marseille; JEAN MICHEL VITON, Principal Investigator — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Cotinat M, Boquet I, Ursino M, Brocard C, Jouve E, Alberti C, Bensoussan L, Viton JM, Brocard F, Blin O. Riluzole for treating spasticity in patients with chronic traumatic spinal cord injury: Study protocol in the phase ib/iib adaptive multicenter randomized controlled RILUSCI trial. PLoS One. 2023 Jan 20;18(1):e0276892. doi: 10.1371/journal.pone.0276892. eCollection 2023. PMID 36662869